CLINICAL TRIAL: NCT04182594
Title: A Phase-II, Randomized, Assessor-Blind, Controlled Trial Comparing the Occurrence of Cardiovascular Events in Patients With Prostate Cancer and Cardiovascular Risk Factors Receiving Degarelix or GnRH Agonist
Brief Title: Cardiovascular Events in GnRH Agonist vs. Antagonist
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0670-19-RMC
Record Dates: First submitted 2019-10-24; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-10

CONDITIONS: Hormone Sensitive Prostate Cancer; Prostate Cancer; Cardiac Event
MeSH Terms: conditions — Prostatic Neoplasms; Cardiovascular Diseases | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Degarelix (Experimental): GnRH Antagonist
  Interventions: Drug: Degarelix
- GnRH-agonist (Active Comparator): GnRH Agonist
  Interventions: Drug: GnRH agonist

INTERVENTIONS:
Drug: Degarelix — Treatment will start with two injections of 120 mg each followed by maintenance of a single injection of 80 mg administered every 28 days
  Other Names: Firmagon
  Arms: Degarelix
Drug: GnRH agonist — GnRH agonist at the discretion of the treating Urologist/Oncologist for 1 year
  Arms: GnRH-agonist

SUMMARY:
The purpose of this study is to test if the use of Degarelix for 1 year associated with a lower rate of cardiovascular toxicity compared to Gonadotropin-releasing hormone (GnRH) agonists in patients with advanced prostate cancer and cardiovascular risk factors, receiving combination therapy of Androgen deprivation therapy (ADT) and second line hormonal or chemotherapy?

DETAILED DESCRIPTION:
Study design: Randomized phase-2, open label superiority study of the use of ADT combined with second line hormonal or chemotherapy in men with advanced prostate cancer and pre-existing cardiovascular risks.

Study population: Subjects with pre-existing cardiovascular risk with locally advanced or metastatic prostate cancer and scheduled to start ADT in combination with either second line hormonal or chemotherapy. We will exclude patients with use of ADT 6 months prior to randomization.

Intervention- Two initial loading doses of 120mg Degarelix for 1 month followed by 80mg monthly for eleven additional months.

Control- GnRH agonist at the discretion of the treating Urologist/Oncologist for 1 year.

Study Time line- The intervention phase will be for one year. During this year, follow-up visits will occur every 3 months. At each visit, we will assess the occurrence of cardiac-related events. In addition, Protein-specific Antigen (PSA) test will be performed each visit. At baseline, 3, 6 and 12 months cardiac biomarkers and lab measurements will be taken. Echocardiogram will be performed at baseline, 6, 9 and 12 months. In addition, cardio-vascular related events and hospitalizations will be monitored for additional 5 years.

Primary endpoint: To compare time to first cardiovascular event of patients with advanced prostate cancer treated for one year with Degarelix vs. GnRH agonist. This will be a composite outcome composed of: Death, Cerebrovascular accident (CVA), Myocardial infarction (MI), Transient ischemic attack (TIA), cardiac emergency room visits, heart catheterization.

Secondary endpoints: To compare time to first major adverse cardiovascular and cerebrovascular event (MACCE)- (Death, CVA, MI, heart catheterization with stent) as estimated by the cumulated probability at the 1-year timepoint of patients with advanced prostate cancer treated for one year with Degarelix vs. LHRH agonist. To compare cardiovascular biomarker levels of patients with advanced prostate cancer treated with Degarelix vs. GnRH agonist. To compare change in cardiac function as measured by Echocardiography in 6,9 and 12 months.

Study impact- This study has the potential to cause a paradigm shift. If we indeed demonstrate that Degarelix is associated with less cardiovascular toxicity with clinical significance, we expect that most urologist, as well as patients, will prefer Degarelix over all other ADT.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced high-risk prostate cancer OR metastatic prostate cancer patients.
2. Patients are scheduled to receive a combination of either

   1. primary ADT for 12 months + either chemotherapy with docetaxel OR
   2. primary ADT for 12 months + second line hormonal treatment with abiraterone/ enzalutamide/ apalutamide
3. Patients with a medical history of either of the following:

   1. Myocardial infarction
   2. Ischaemic or haemorrhagic cerebrovascular conditions
   3. Arterial embolic and thrombotic events
   4. Ischaemic heart disease
   5. Prior coronary artery or iliofemoral artery revascularization (percutaneous or surgical procedures)
   6. Peripheral vascular disease (e.g. significant stenosis (ABPI<0.9), claudication, prior vascular surgery/intervention(
   7. Two out of three cardiovascular risk factors: hypertension, diabetes, current smoking.
4. Patients age 18-90 years.
5. Life expectancy of over 12 months.
6. WHO performance status of 0-2
7. Subject is able and has agreed to sign a consent form.

Exclusion Criteria:

1. Prior use of ADT in past 6 months prior to randomization. We will, however, allow prior use of anti-androgens such as Casodex, Chimax, Drogenil, and Cyprostat.
2. Known allergic reaction to Degarelix.
3. Any psychological, familial, sociological or geographical situation potentially hampering compliance with the study protocol and follow-up schedule.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-17 (Estimated); Primary Completion 2023-01-17 (Estimated); Study Completion 2023-01-17 (Estimated)

PRIMARY OUTCOMES:
time to first cardiovascular event | 1 year
  To compare time to first cardiovascular event as estimated by the cumulated probability at the 1-year time-point of patients with advanced prostate cancer treated for one year with Degarelix vs. GnRH agonist. This will be a composite outcome composed of: Death, CVA, MI, TIA, cardiac emergency room visits, heart catheterization.

SECONDARY OUTCOMES:
time to first MACCE event | 1 year
  To compare time to first MACCE event as estimated by the cumulated probability at the 1-year timepoint of patients with advanced prostate cancer treated with Degarelix vs. GnRH agonist and combination therapy.
  MACCE will be defined as:
  1. Death of any cause
  2. MI
  3. CVA
  4. Percutaneous coronary intervention, (PCI) with stent insertion
cardiac echocardiography | 1 year
  To compare change in ejection fraction (EF) as measured by cardiac echocardiography of patients with advanced prostate cancer treated with Degarelix vs. GnRH agonist, at baseline, six-, nine- and twelve-months of combination treatment.
Hormonal Profile | 1 year
  To compare testosterone serum levels (ng/dL) of patients with advanced prostate cancer treated with Degarelix vs. GnRH agonist, at baseline, three-, six- and twelve-months of combination treatment.
NTproBNP levels | 1 year
  To compare levels of NTproBNP (pg/mL) in patients with advanced prostate cancer treated with Degarelix vs. GnRH agonist, at baseline, three-, six-, nine- and twelve-months of combination treatment.
Adverse events | 1 year
  To compare rate of other adverse events in patients with advanced prostate cancer treated with Degarelix vs GnRH agonist and combination therapy.
PSA levles | 1 year
  To compare PSA serum levels (ng/mL) of patients with advanced prostate cancer treated with Degarelix vs. GnRH agonist, at baseline, three-, six- nine- and twelve-months of combination treatment.
BMI | 1 year
  To compare changes in body mass index (BMI) in patients with advanced prostate cancer treated with Degarelix vs. GnRH agonist, at baseline, three-, six- and twelve-months of combination treatment.
Quality of life: FACT-P questionnaire | 1 year
  To compare the quality of life by self-reported FACT-P questionnaire, by patients with advanced prostate cancer treated with Degarelix vs. GnRH agonist, at baseline, three-, six- and twelve-months of combination treatment
Glucose profile | 1 year
  To compare glucose levels (mg/dL) in patients with advanced prostate cancer treated with Degarelix vs GnRH agonist, at baseline, three-, six- and twelve-months of combination treatment.
Cholesterol levles | 1 year
  To compare Cholesterol serum levels (mg/dL) of patients with advanced prostate cancer treated with Degarelix vs. GnRH agonist, at baseline, three-, six- nine- and twelve-months of combination treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD, PhD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center - Beilinson Hospital, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976